CLINICAL TRIAL: NCT03571412
Title: Comparative of Antidepressive Effect on 5Hz rTMS on Dorsomedial Prefrontal Cortex and Left Dorsolateral Prefrontal Cortex
Brief Title: Antidepressive Effect on 5 Herz (Hz) rTMS Over Dorsomedial Prefrontal Cortex and Left Dorsolateral Prefrontal Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Queretaro (Other)
Responsible Party: Principal Investigator, Dr. Julian Reyes López, Professor, Universidad Autonoma de Queretaro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-05/05/2016
Record Dates: First submitted 2018-01-10; First posted 2018-06-27 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The purpose to this study is to valuate the clinical effects of 5Hz rTMS over Left Dorsolateral Prefrontal Cortex and Dorsomedial Prefrontal Cortex
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5Hz Left Dorsolateral Prefrontal Cortex (Experimental): This group will receive 5Hz Left Dorsolateral Prefrontal Cortex repetitive Transcranial Magnetic Stimulation. Once a day on monday to friday. Until complete 15 sessions.After complete acute phase intervention (15 sessions) subject will have a 5 week clinical follow up.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- 5Hz Dorsomedial Prefrontal Cortex (Experimental): This group will receive 5Hz Dorsomedial Prefrontal Cortex Transcranial Magnetic Stimulation, once a day on monday to friday. Until complete 15 sessions.After complete acute phase intervention (15 sessions) subject will have a 5 week clinical follow up.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — Subject will receive 5Hz LDLPFC or 5Hz DMPFC rTMS
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
This study evaluates the efficacy of 5Hz repetitive Transcranial Magnetic Stimulation (rTMS) over Left Dorsolateral Prefrontal Cortex and Dorsomedial Prefrontal Cortex on Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) affects a significant percentage of the national population (17-20%) in 2:1 ratio in women compared to men. Repetitive Transcranial Magnetic Stimulation (rTMS) is an effective neuromodulation technique for the treatment of Major Depressive Disorder and it has demonstrated favorable clinical effects when applied over the Left Dorsolateral Prefrontal Cortex (LDLPFC); however there is evidence that other areas of the prefrontal cortex such as the Dorsomedial Prefrontal Cortex (DMPFC) could be ideal for rTMS treatment targets during the presence of MDD, given its association with deficient cognitive processes during the course of the illness. There is also evidence of the use of 5Hz frequency with the same clinical effectiveness from other frequencies such as 10 Hz and 20 Hz when applied to the LDLPFC. However, there are no current research that have addressed the use of this frequency on DMPFC.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old.
* Meet DSM 5 (Diagnostic and Statistical Manual, 5 edition) diagnostic criteria for Major Depressive Disorder.
* Score >17 in Hamilton Depression Rating Scale.

Exclusion Criteria:

* Subjects with diagnose of Psychotic Depression, Schizophrenia, Bipolar Disorder, Post Traumatic Stress Disorder.
* Subjects with epilepsy or presence of paroxysms during the EEG.
* Subjects with previous history of traumatic brain injury, metal plates in the skull, cochlear devices, infusion devices such as insulin pumps.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms evaluated by Hamilton Depressive Rating Scale (HADRS) | 3 weeks
  Hamilton Depressive Rating Scale (HADRS) is a 21 item clinimetric scale to evaluate severity of depressive symptoms in patients.

SECONDARY OUTCOMES:
Changes in depressive symptoms evaluated by Montgomery-Asberg Depressive Rating Scale (MADRS) | 3 weeks
  Montgomery- Asberg Depressive Rating Scale (MADRS) is a 10 item clinimetric scale that evaluates the presence and severity of depressive symptoms in subjects with the disorder mentioned before.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Reyes, PhD, Study Director — Universidad Autónoma de Querétaro